CLINICAL TRIAL: NCT04825613
Title: "Individual Patient Expanded Access IND to Evaluate the Safety and Efficacy of HB-adMSCs for the Treatment of Primary Lateral Sclerosis"
Brief Title: "Individual Patient Expanded Access IND to Treat Primary Lateral Sclerosis"
Status: No longer available | Type: Expanded Access
Sponsor: Hope Biosciences Research Foundation (Industry)
Responsible Party: Sponsor
Other Study IDs: HBPLS01
Record Dates: First submitted 2021-03-25; First posted 2021-04-01 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Primary Lateral Sclerosis, Adult, 1
Keywords: Primary Lateral Sclerosis, PLS, Sclerosis
MeSH Terms: conditions — Primary Lateral Sclerosis, Adult, 1; Motor Neuron Disease; Papillon-Lefevre Disease; Sclerosis

INTERVENTIONS:
Biological: HB-adMSCs — Hope Biosciences adipose derived Mesenchymal Stem Cells
  Other Names: MSC's

SUMMARY:
This Individual Patient Expanded Access IND has been created as requested by an 83-year-old man who suffers Primary Lateral Sclerosis and for which the drugs currently approved are not providing an improvement over the progression of this disease.

DETAILED DESCRIPTION:
-Screening This expanded access IND was created at the request of the subject who already has his own stem cells banked at Hope Biosciences, LLC. After receiving authorization from FDA and Western IRB, the subject will be contacted and provided with a copy of the informed consent for review. The Principal Investigator or delegated staff will meet with the patient in person or by telephone and explain the study procedures (including cell infusion, and safety assessment procedures), follow-up visits, potential risks and benefits of the study, alternatives, and the voluntary nature of participation.

Ample time will be given for the patient to ask questions and make a decision about participation. If consent is obtained, the principal investigator or delegated staff will collect patient's medical history and schedule the date for the Infusion 1. The informed consent process will be documented in the subject's record and will include the discussion points mentioned above. A copy of the signed informed consent will be placed in the record.

-HB-adMSCs Administrations. Subject will receive a total of twelve autologous HB-adMSCs infusion of 200 million cells with a dosing interval of 28 days over a 44-week period during the first and second year of treatment. Laboratory assessments will be collected at different visits across the study.

Other assessments should be completed during these visits by the Investigator and/or delegated staff to evaluate the safety and efficacy of HB-adMSCs,

1. Collection of Medical History
2. Collection of Concomitant Medications.
3. Collection of Vital Signs (Respiratory Rate, Blood Pressure, Body Temperature, Heart Rate and Oxygen Saturation). Vital Signs will be collected for 2 hours post investigational product exposure. Every 15 minutes for the first hour and every 30 minutes after that. If it is indicated by principal investigator vital signs should be collected more frequently.
4. Collection of Weight and Height (Height measurement is only necessary at infusion 1)
5. EMG NCV is required to be completed at Infusion 1 and 7. If an EMG NCV has not been done within 28 days of these visit, the Principal Investigator will place an order to obtain it. Any EMG NCV done within 28 days of the visit as standard of care can be used for this requirement.
6. Physical Examination.
7. ALS Functional Rating Scale-Revised (ALSFRS-R) at Infusion 1 and 7.
8. Neuro QOL Scale at Infusion 1 and 7.
9. A video documentation of the subject will be recorded during Infusion 1 and 7 with the purpose of observing his usual forms of communication and movements.
10. Laboratory Samples. A blood sample for clinical labs - CBC with Platelets, CMP, PT, PTT, INR, as well as C-reactive protein, Sedimentation Rate and Vitamin B12 (Cobalamin) to be collected at Infusion 1 and 7.
11. Telephone Encounter 24 hours after each infusion to evaluate the incidence of any Adverse event or Serious Adverse Events.

    * Follow Up 1 Week 48. (Phone call)

1. Update medical history and concomitant medications if there is any new information.

2. Assess the incidence of any Adverse event or Serious Adverse Events since last infusion.

* Infusions 13 through 24.

  1. Collection of Medical History
  2. Collection of Concomitant Medications.
  3. Collection of Vital Signs (Respiratory Rate, Blood Pressure, Body Temperature, Heart Rate and Oxygen Saturation). Vital Signs will be collected for 2 hours post investigational product exposure. Every 15 minutes for the first hour and every 30 minutes after that. If it is indicated by principal investigator vital signs should be collected more frequently.
  4. Collection of Weight and Height (Height measurement is only necessary at infusion 1)
  5. EMG NCV is required to be completed at Infusion 13 and 19. If an EMG NCV has not been done within 28 days of these visit, the Investigator will place an order to obtain it.

     Any EMG NCV done within 28 days of the visit as standard of care can be used for this requirement.
  6. Physical Examination.
  7. ALS Functional Rating Scale-Revised (ALSFRS-R) at Infusion 13 and 19.
  8. Neuro QOL Scale at Infusion 13 and 19.
  9. A video documentation of the subject will be recorded during Infusion 13 and 19 with the purpose of observing his usual forms of communication and movements.
  10. Laboratory Samples. A blood sample for clinical labs - CBC with Platelets, CMP, PT, PTT, INR, as well as C-reactive protein, Sedimentation Rate and Vitamin B12 (Cobalamin) to be collected at Infusion 13 and 19.
  11. Telephone Encounter 24 hours after each infusion to evaluate the incidence of any Adverse event or Serious Adverse Events.
* End of Study (Week 52)

  1. Update medical history and concomitant medications if there is any new information.
  2. Assess the incidence of any Adverse Event or Serious Adverse Events since last visit.
  3. Collection of Weight.
  4. Collection of Vital Signs (Respiratory Rate, Blood Pressure, Body Temperature, Heart Rate and Oxygen Saturation).
  5. Laboratory Samples. A blood sample for clinical labs - CBC with Platelets, CMP, PT, PTT, INR, as well as C-reactive protein, Sedimentation Rate and Vitamin B12 (Cobalamin).
  6. Physical Examination.
  7. ALS Functional Rating Scale-Revised (ALSFRS-R).
  8. Neuro QOL Scale.
  9. A video documentation of the subject will be recorded during this visit with the purpose of observing his usual forms of communication and movements.
  10. EMG NCV is required to be completed at EOS visit. If an EMG NCV has not been done within 28 days of this visit, the Principal Investigator will place an order to obtain it. Any EMG NCV done within 28 days of the visit as standard of care can be used for this requirement.

ELIGIBILITY:
HBPLS01

Inclusion Criteria:

1. Adult individual at least 18 years old
2. Clinical diagnosis Primary Lateral Sclerosis.
3. Subject or Legal Authorized Representative has provided informed consent before initiation of any study procedure.
4. Subject has mesenchymal stem cells banked at Hope Biosciences.

Exclusion Criteria:

1. Clinically significant, uncontrolled cardiovascular, lung, renal, hepatic, or endocrine disease or any other acute or chronic medical condition that, in the opinion of the principal investigator, may increase the risks associated with study participation.
2. Chemical or ETOH dependency that in the opinion of the investigator would preclude participation in the study.
3. Participation in concurrent interventional research studies during this expanded access.
4. Unwillingness to return for follow-up visits.

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Djamchid Lotfi, MD, Principal Investigator — Hope Biosciences Stem Cell Research Foundation
Locations (1):
- Hope Biosciences Stem Cell Research Foundation, Sugar Land, Texas, United States